CLINICAL TRIAL: NCT00628368
Title: Study to Analyze the Predictive Role of Factors Implicated in the Signaling Pathway of the EGFR in Response to Treatment With Neoadjuvant Chemoradiotherapy in Patients With Cancer of the Esophagus or Rectum
Brief Title: Biological Factors in Predicting Response to Treatment in Patients With Esophageal Cancer or Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000574175; CLCC-EGFR-BIO; INCA-RECF0366
Record Dates: First submitted 2008-03-01; First posted 2008-03-05 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; adenocarcinoma of the rectum; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Rectal Neoplasms | interventions — Gene Expression Profiling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Rectal and oesophagus cancer (Experimental): Additionnal samples from routine care (tumor tissue and healthy tissue and one blood tube) and standardized clinical data will be entered into a database.
  Interventions: Genetic: Gene expression analysis

INTERVENTIONS:
Genetic: Gene expression analysis — Tissue samples (tumor tissue and healthy tissue) frozen and secured in paraffin collected during surgery. One blood tube will be frozen.
  During a coloscopy or gastroscopy tumor and health tissue samples will be taken for diagnosis and research.

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying how well biological factors work in predicting response to treatment in patients with esophageal cancer or rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Analyze various biological factors that can be used as markers to predict response to treatment and correlate with the signaling pathway of EGFR.

Secondary

* Establish a tissue bank to store information about the response to treatment and survival.

OUTLINE: Patients undergo endoscopy, 11 biopsies of tumor tissue, and 3 biopsies of healthy mucosa. Blood samples are also collected. Samples are analyzed for the expression of 4 receptors in the EGFR family, polymorphisms at intron 1 of the EGFR gene, and gene mutations in downstream signaling pathways.

After surgery, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus or rectum
* Planning to receive neoadjuvant treatment, including radiotherapy or chemoradiotherapy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* No blood disorder
* Not deprived of freedom or protected by law

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09-30 (Actual)

PRIMARY OUTCOMES:
Determination of predictive factors in the EGFR signaling pathway in response to treatment | End of study : approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Result] Arsic N, Ho-Pun-Cheung A, Lopez-Crapez E, Assenat E, Jarlier M, Anguille C, Colard M, Pezet M, Roux P, Gadea G. The p53 isoform delta133p53ss regulates cancer cell apoptosis in a RhoB-dependent manner. PLoS One. 2017 Feb 17;12(2):e0172125. doi: 10.1371/journal.pone.0172125. eCollection 2017. PMID 28212429